CLINICAL TRIAL: NCT00275002
Title: A Phase II Trial of O6-Benzylguanine and Temozolomide in Pediatric Patients With Recurrent or Progressive High-Grade Gliomas and Recurrent or Progressive Brainstem Tumors
Brief Title: O6-Benzylguanine and Temozolomide in Treating Young Patients With Recurrent or Progressive Gliomas or Brain Stem Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03050; PBTC-015; NCI-06-C-0089; NCI-P6692; CDR0000455561 (Registry Identifier: PDQ (Physician Data Query)); NCT00291291 (obsolete NCT alias)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent childhood brain stem glioma; recurrent childhood brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — O(6)-benzylguanine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- O6-BG and TMZ (Experimental): O6-benzylguanine (O6-BG) and temozolomide (TMZ)
  Interventions: Drug: O6-benzylguanine; Drug: temozolomide

INTERVENTIONS:
Drug: O6-benzylguanine — Dosing is based on the body surface area (BSA) calculated at the beginning of each course of therapy. O6-Benzylguanine, 120 mg/m^2, will be administered as a one-hour intravenous (IV) infusion, daily for 5 days. Four consecutive weeks will constitute one course. Courses will be repeated every 4 weeks for up to 12 courses of therapy.
Drug: temozolomide — Dosing is based on the body surface area (BSA) calculated at the beginning of each course of therapy. Temozolomide, 75 mg/m^2 (rounded to the nearest 5 mg, the size of the smallest capsule) will be given orally, 30 minutes following the completion of each infusion of O6-Benzylguanine. Four consecutive weeks will constitute one course. Courses will be repeated every 4 weeks for up to 12 courses.
  Other Names: Temodar

SUMMARY:
This phase II trial is studying how well giving O6-benzylguanine together with temozolomide works in treating young patients with recurrent or progressive gliomas or brain stem tumors. Drugs used in chemotherapy, such as O6-benzylguanine and temozolomide , work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. O6-benzylguanine may help temozolomide work better by making tumor cells more sensitive to the drug. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the sustained objective response rate to the combination of O6-benzylguanine and temozolomide in pediatric patients with recurrent or progressive high-grade gliomas and brain stem tumors.

SECONDARY OBJECTIVES:

I. Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to tumor type (high-grade gliomas vs brain stem tumors).

Patients receive O6-benzylguanine IV over 1 hour followed by oral temozolomide on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed to the earliest of 30 days following discontinuation of therapy or the initiation of additional anti-cancer therapy or death.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA

* Tumor: Participants must have a high-grade glioma (including e.g. histologically confirmed anaplastic astrocytoma, glioblastoma multiforme, anaplastic oligodendroglioma, anaplastic ganglioma, gliosarcoma) or a brainstem tumor (histologic confirmation waived) with documentation of disease recurrence or progression after treatment with standard therapy. Participants must have bi-dimensionally measurable disease, defined as at least 1 lesion that can be measured in ≥ 2 dimensions
* Age: 21 years of age or less
* Performance status: Karnofsky 60-100% (for patients > 16 years of age) or Lansky 60-100% (for patients ≤ 16 years of age)
* Life expectancy: Not specified
* Hematopoietic: Must have adequate bone marrow function defined as absolute neutrophil count > 1,500/mm^3, platelet count > 100,000/mm^3 (unsupported), hemoglobin > 8 g/dL (may be supported), and absolute lymphocyte count ≥ 500/mm^3
* Hepatic: Must have SGOT and SGPT ≤ 2.5 times upper limit of normal (ULN), bilirubin ≤ 1.5 times ULN, and no overt hepatic disease
* Renal: Participants must have creatinine clearance ≥ 60 mL/min or creatinine based on age as follows: no greater than 0.8 mg/dL (for patients ≤ 5 years of age), no greater than 1.0 mg/dL (for patients 6 to 10 years of age), no greater than 1.2 mg/dL (for patients 11 to 15 years of age), or no greater than 1.5 mg/dL (for patients > 15 years of age). There must be no overt renal disease
* Cardiovascular: Must have no overt cardiac disease
* Pulmonary: Must have no overt pulmonary disease
* Other: Female participants of childbearing potential must have a negative pregnancy test prior to study registration, and must avoid breast-feeding. Female and male participants of childbearing or child-fathering potential must use effective contraception
* Bone Marrow Transplant: Must be at least 6 months since prior allogeneic bone marrow transplantation and at least 3 months since prior autologous bone marrow or stem cell transplantation
* Growth Factors: Must be at least 2 weeks since prior colony-stimulating factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF], or erythropoietin)
* Prior Chemotherapy: Must have received last dose of myelosuppressive anticancer chemotherapy ≥ 3 weeks prior to study registration and ≥ 6 weeks for nitrosoureas. Must have received last dose of nonmyelosuppressive investigational agents or anticancer drugs ≥ 7 days prior to study registration. Participants who have received prior temozolomide are eligible
* Concurrent Endocrine Therapy: Concurrent corticosteroid therapy is allowed
* Prior Radiotherapy: Must have received last fraction of craniospinal irradiation and local irradiation to the primary tumor ≥ 12 weeks prior to study registration
* Prior Therapy-Other: Must have recovered from all prior therapy

EXCLUSION CRITERIA

* Must not have history of severe toxicity (≥ grade 3) associated with temozolomide
* Must not be receiving other concurrent anticancer or investigational therapy
* Must not have history of hypersensitivity to dacarbazine, temozolomide, or polyethylene glycol (PEG)
* Must not have uncontrolled significant systemic illness including infection, or overt renal, hepatic, cardiac, or pulmonary disease
* Must not be HIV positive

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2006-02; Primary Completion 2010-12-01 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Warren, MD, Study Chair — National Cancer Institute (NCI)
Locations (11):
- United States (11):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas
  - Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from PBTC member institutions were enrolled between October 2005 and February 2008.
Groups:
- Recurrent High-Grade Gliomas: Participants with recurrent or progressive high-grade gliomas receive 120 mg/m^2 of O6-Benzylguanine administered as a one-hour intravenous infusion, daily for 5 days. Temozolomide, 75 mg/m^2 is administered orally, 30 minutes following the completion of each infusion of O6-Benzylguanine. Four consecutive weeks will constitute one course, and courses will be repeated every 4 weeks.
- Recurrent Brain Stem Tumors: Participants with recurrent or progressive brain stem tumors receive 120 mg/m^2 of O6-Benzylguanine administered as a one-hour intravenous infusion, daily for 5 days. Temozolomide, 75 mg/m^2 is administered orally, 30 minutes following the completion of each infusion of O6-Benzylguanine. Four consecutive weeks will constitute one course, and courses will be repeated every 4 weeks.
Period: Overall Study
Arm/Group | Recurrent High-Grade Gliomas | Recurrent Brain Stem Tumors
Started | 25 | 16
Completed | 3 | 0
Not Completed | 22 | 16
Not completed — Death | 1 | 0
Not completed — Disease progression | 21 | 15
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recurrent High-Grade Gliomas | Recurrent Brain Stem Tumors | Total
Number analyzed (Participants) | 25 | 16 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 16 | 39
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (5.1) | 7.8 (3.9) | 11.2 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 16 | 4 | 20
Region of Enrollment [Number; unit: participants]
  United States | 25 | 16 | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Objective Response (Complete Response or Partial Response)
Description: The primary endpoint is to assess the percentage of participants with a sustained objective response (complete response (CR) or partial response (PR)). Response is assessed by magnetic resonance imaging (MRI) per the following criteria: CR - disappearance of tumor and PR - ≥50% reduction in tumor based on the maximal cross-sectional measurements. The response must be sustained for at least 8 weeks, and the date of the confirmed sustained response is the date at which the response was first noted by MRI.
Time Frame: Week 8, 16, 24, 32, and 40 after starting therapy
Population: Participants included in assessing objective response were those who completed two courses of therapy or those who died or experienced progressive disease prior to completing the second course.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Recurrent High-Grade Gliomas | Recurrent Brain Stem Tumors
Number analyzed (Participants) | 25 | 16
Percent of Participants | 4 [0.1 to 20] | 0 [0 to 21]

2. Secondary Outcome: Number of Patients With Grade 3 or 4 Adverse Events at Least Possibly Related to the Combination of O6-benzylguanine and Temozolomide
Description: Clinical and laboratory studies to assess adverse events are obtained at least every four weeks (prior to each course) with some laboratory studies obtained every 2 weeks. Adverse events are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0). Attribution of each adverse event to the treatment regimen is determined by the participant's attending physician at the enrolling institution and verified by the study chair.
Time Frame: From day 1 of therapy up to 49 months
Population: Participants who received at least one day of the treatment regimen were included in the analysis of this objective.
Measure: Number; unit: Participants
Arm/Group | Recurrent High-Grade Gliomas | Recurrent Brain Stem Tumors
Number analyzed (Participants) | 25 | 16
Participants | 16 | 10

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from day 1 of starting treatment until 30 days after ceasing treatment (off study). AEs possibly, probably, or definitely attributed to the study drug that occur after the patient is off the study are also collected.
Arm/Group | Recurrent High-Grade Gliomas | Recurrent Brain Stem Tumors
Serious Adverse Events (participants affected / at risk) | 15/25 | 12/16
Other Adverse Events (participants affected / at risk) | 25/25 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Recurrent High-Grade Gliomas (N=25) | Recurrent Brain Stem Tumors (N=16)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Bilirubin (Investigations) | 1 | 0
Colitis, infectious (Infections and infestations) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Leukocytes (total WBC) (Investigations) | 2 | 3
Lipase (Investigations) | 1 | 0
Lymphopenia (Investigations) | 0 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Mental Status (Nervous system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Neutrophils/granulocytes (Investigations) | 6 | 5
Phlebitis (Vascular disorders) | 0 | 1
Platelets (Investigations) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Somnolence (Nervous system disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Recurrent High-Grade Gliomas (N=25) | Recurrent Brain Stem Tumors (N=16)
ALT,SGPT (Investigations) | 6 | 3
ALT,SGOT (Investigations) | 3 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 2
Alkaline phosphatase (Investigations) | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 3 | 0
Ataxia (Nervous system disorders) | 0 | 3
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 3 | 4
Bilirubin (Investigations) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 1
Constipation (Gastrointestinal disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cushingoid appearance (Endocrine disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 5
Dizziness (Nervous system disorders) | 4 | 2
Dry eye syndrome (Eye disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Edema:limb (General disorders) | 0 | 1
Edema:trunk/genital (General disorders) | 0 | 1
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
gamma-Glutamyl transpeptidase (Investigations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 10 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 5 | 3
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 2 | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 | 1
Hemoglobinuria (Renal and urinary disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Injection site reaction/extravasation changes (General disorders) | 0 | 1
Leukocytes (total WBC) (Investigations) | 15 | 9
Lymphopenia (Investigations) | 13 | 8
Hypermagnesemia (Metabolism and nutrition disorders) | 5 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 10 | 4
Neutrophils/granulocytes (Investigations) | 13 | 9
Nystagmus (Nervous system disorders) | 0 | 1
Partial thromboplastin time (Investigations) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 4
Platelets (Investigations) | 16 | 10
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 7 | 4
Proteinuria (Renal and urinary disorders) | 0 | 1
Pyramidal tract dysfunction (Nervous system disorders) | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 4 | 2
Tremor (Nervous system disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 11 | 7
Weight loss (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less